CLINICAL TRIAL: NCT00004857
Title: A Phase II Study of Fludarabine Induction Followed by CAMPATH-1H Consolidation in Untreated Patients With B-Cell Chronic Lymphocytic Leukemia
Brief Title: Fludarabine Followed by Alemtuzumab in Treating Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-19901; U10CA031946 (NIH); CDR0000067506 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2000-03-07; First posted 2003-12-11 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Leukemia
Keywords: stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fludarabine + Campath-1H (Experimental): Standard of care induction with fludarabine followed by consolidation antibody therapy
  Interventions: Biological: alemtuzumab; Drug: fludarabine phosphate

INTERVENTIONS:
Biological: alemtuzumab — 30 mg subQ injection tiw for 6 weeks
  Other Names: campath-1H
Drug: fludarabine phosphate — 25mg/sq m/day IV infusion x 5 days Wks 1, 5, 9, and 13

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as alemtuzumab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells.

PURPOSE: Phase II trial to study the effectiveness of fludarabine followed by alemtuzumab in treating patients who have chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the overall response rate of previously untreated patients with stage I, II, III, or IV B-cell chronic lymphocytic leukemia when treated with fludarabine induction followed by alemtuzumab consolidation. II. Determine the infectious toxic effects and feasibility of this regimen in this patient population. III. Determine the treatment-related toxic effects, including infection and injection site reactions, of subcutaneous vs intravenous alemtuzumab in patients treated with this regimen. IV. Determine the progression-free and overall survival of patients treated with this regimen. V. Determine the immunologic effects of this regimen in these patients.

OUTLINE: Patients receive fludarabine IV over 30 minutes 5 days a week. Treatment repeats every 28 days for 4 courses in the absence of disease progression. Patients undergo clinical staging after completion of course 4 of fludarabine followed by 2 months of observation. Patients with stable or responding disease receive alemtuzumab subcutaneously 3 days a week for 6 weeks. Patients undergo clinical staging again after completion of 6 weeks of alemtuzumab followed by 2 more months of observation. Patients are followed every 3 months for 1 year and then every 6 months for 8 years.

ELIGIBILITY:
1. Specific Diagnosis of B-Cell CLL

   1.1 An absolute lymphocytosis of > 5,000/µl

   1.1.1 Morphologically, the lymphocytes must appear mature with < 55% prolymphocytes.

   1.1.2 Bone marrow examination must include at least a unilateral aspirate and biopsy. The aspirate smear must show > 30% of all nucleated cells to be lymphoid or the bone marrow core biopsy must show lymphoid infiltrates compatible with marrow involvement by CLL. The overall cellularity must be normocellular or hypercellular.

   1.1.3 Local institution lymphocyte phenotype must reveal a predominant B-cell monoclonal population sharing a B-cell marker (CD19, CD20, CD23, CD24) with the CD5 antigen, in the absence of other pan-T-cell markers. Additionally, the B-cells must be monoclonal with regard to expression of either κ or λ and have surface immunoglobulin expression of low density. Patients with bright surface immunoglobulin levels must have CD23 co-expression.

   1.2 Staging

   1.2.1 Patients must be in the intermediate- or high-risk categories of the modified three-stage Rai staging system (i.e., stages I, II, III, or IV) per the protocol.

   1.2.2 Patients in the intermediate-risk group must have evidence of active disease as demonstrated by at least one of the following criteria:
   * Massive or progressive splenomegaly and/or lymphadenopathy
   * Presence of weight loss > 10% over the preceding 6 month period;
   * Grade 2 or 3 fatigue
   * Fevers > 100.5°C or night sweats for greater than 2 weeks without evidence of infection
   * Progressive lymphocytosis with an increase of > 50% over a 2 month period or an anticipated doubling time of less than 6 months.
2. Prior Treatment: No prior therapy for CLL including corticosteroids for autoimmune complications that have developed since the initial diagnosis of CLL.
3. No medical condition requiring chronic use of oral corticosteroids.
4. Age ≥18 years.
5. Performance Status 0 - 2.
6. No HIV disease. Due to alterations in host immunity, patients with HIV may not be enrolled.
7. Non-pregnant and non-nursing. Due to the unknown teratogenic potential of Campath-1H, pregnant or nursing women may not be enrolled. Women and men of reproductive potential should agree to use an effective means of birth control.
8. Initial Required Laboratory Values:

Creatinine <1.5 x upper limit of institutional normal value Coomb's Testing NEGATIVE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2000-01; Primary Completion 2003-03 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Response | 2 months post consolidation

SECONDARY OUTCOMES:
Toxicity | 2 months post consolidation

CONTACTS AND LOCATIONS:
Overall Officials: Kanti R. Rai, MD, Study Chair — Long Island Jewish Medical Center
Locations (50):
- United States (50):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - CCOP - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Background] Morrison VA, Peterson BL, Rai KR, et al.: Alemtuzumab increases serious infections in patients with previously untreated chronic lymphocytic leukemia (CLL) receiving fludarabine-based therapy: a comparative analysis of 3 Cancer and Leukemia Group B studies (CALGB 9011, 9712, 19901). [Abstract] Blood 110 (11): A-756, 2007.
- [Background] Rai KR, Freter CE, Mercier RJ, Cooper MR, Mitchell BS, Stadtmauer EA, Santabarbara P, Wacker B, Brettman L. Alemtuzumab in previously treated chronic lymphocytic leukemia patients who also had received fludarabine. J Clin Oncol. 2002 Sep 15;20(18):3891-7. doi: 10.1200/JCO.2002.06.119. PMID 12228210
- [Result] Byrd JC, Peterson BL, Rai KR, Hurd D, Hohl R, Perry MC, Gockerman J, Nattam S, Larson RA. Fludarabine followed by alemtuzumab consolidation for previously untreated chronic lymphocytic leukemia: final report of Cancer and Leukemia Group B study 19901. Leuk Lymphoma. 2009 Oct;50(10):1589-96. doi: 10.1080/10428190903150839. PMID 19863336
- [Result] Rai KR, Byrd JC, Peterson B: Subcutaneous alemtuzumab following fludarabine for previously untreated patients with chronic lymphocytic leukemia (CLL): CALGB study 19901. [Abstract] Blood 102 (11 Pt 1): A-2506, 2003.
- [Result] Rai KR, Byrd JC, Peterson BL, et al.: A phase II trial of fludarabine followed by alemtuzumab (Campath-1H) in previously untreated chronic lymphocytic leukemia (CLL) patients with active disease: Cancer and Leukemia Group B (CALGB) study 19901. [Abstract] Blood 100 (11 Pt 1): A-772, 2002.
- [Derived] Jones JA, Ruppert AS, Zhao W, Lin TS, Rai K, Peterson B, Larson RA, Marcucci G, Heerema NA, Byrd JC. Patients with chronic lymphocytic leukemia with high-risk genomic features have inferior outcome on successive Cancer and Leukemia Group B trials with alemtuzumab consolidation: subgroup analysis from CALGB 19901 and CALGB 10101. Leuk Lymphoma. 2013 Dec;54(12):2654-9. doi: 10.3109/10428194.2013.788179. Epub 2013 May 9. PMID 23547837